CLINICAL TRIAL: NCT03471468
Title: Study of the Kinetics of Microparticles Under Chemotherapy in Patients With Gastric or Pancreatic Cancer
Brief Title: Kinetics of Microparticles Under Chemotherapy in Patients With Gastric or Pancreatic Cancer
Acronym: DOMICA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DOMICA
Record Dates: First submitted 2018-02-12; First posted 2018-03-20 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Pancreatic Cancer; Gastric Cancer
Keywords: Microparticles; Pancreatic cancer; Gastric cancer; Chemotherapy; Venous thromboembolism
MeSH Terms: conditions — Pancreatic Neoplasms; Stomach Neoplasms; Venous Thromboembolism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- kinetics of microparticles under chemotherapy (Experimental): kinetics of microparticles under chemotherapy in patients with pancreatic or gastric cancer by serial measurements of microparticles procoagulant activity.
  Interventions: Procedure: kinetics of microparticles under chemotherapy

INTERVENTIONS:
Procedure: kinetics of microparticles under chemotherapy — Blood samples done before chemotherapy and 6 hours later for each of six chemotherapies required by the protocol.

SUMMARY:
Microparticles have recently emerged as a thrombotic risk marker with a potential role in determining which patients are at greatest risk for developing thrombosis. Available data show an increase in the level of microparticles in cancer patients who are undergoing chemotherapy for solid tumors with a possible link to their thrombogenic state.

Our study focuses on the kinetics of microparticles under chemotherapy in patients with pancreatic or gastric cancer by serial measurements of microparticles procoagulant activity.

Detailed Description:

The impact of chemotherapy on microparticles expression will be assessed by measuring their procoagulant activity on blood samples taken during the course of chemotherapy. The thrombotic risk will be evaluated by the score of Khorana in parallel. Microparticles expression in patients with thrombosis will be compared to that in other patients.

ELIGIBILITY:
Inclusion Criteria:

* First-line chemotherapy indicated and accepted by the patient for pancreatic cancer or gastric cancer
* Confirmed diagnosis of pancreatic cancer or gastric cancer
* Free subject, without guardianship or trusteeship or subordination
* Patient benefiting from a social security scheme or benefiting through a third party
* Consent given by the patient after clear and fair information about the study

Exclusion Criteria:

* Age < 18yo
* Life expectancy ≤10days
* Deep vein thrombosis ou pulmonary embolism ≤3months
* Patient unable to receive chemotherapy (sepsis, acute coronary syndrome, recent stroke, heparin-induced thrombocytopenia, disseminated intravascular coagulation)
* Person enjoying enhanced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social institution, adults under legal protection, and finally patients in emergency situations
* Pregnant or lactating woman and woman of childbearing age lacking effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Microparticles level will be assessed by automated and standardised measure of their procoagulant power using Kit STA©Procoag-PPL (Diagnostica Stago, Asnière, France) | Before chemotherapies #1 to #6
Microparticles level will be assessed by automated and standardised measure of their procoagulant power using Kit STA©Procoag-PPL (Diagnostica Stago, Asnière, France) | After 6 hours of chemotherapies #1 to #6

SECONDARY OUTCOMES:
incidence of thrombosis during study | Before chemotherapies #1 to #6 and one year after inclusion.
  Deep vein thrombosis or pulmonary embolism
Khorana score does assess the risk of thrombosis uner chemotherapy according to 3 levels :Score 0, 1, 2 or 3 | Before chemotherapies #1 to #6
  Score 0= low risk (incidence of thrombosis = 0.3%) Score 1 or 2= intermediate risk (incidence of thrombosis = 2%) Score >3 = high risk (incidence of thrombosis = 6.7%) The highest possible score is 6.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No